CLINICAL TRIAL: NCT01595386
Title: Effect of Postoperative Hydrocortisone on Cardiovascular and Respiratory Function in Neonates Undergoing Cardiopulmonary Bypass
Brief Title: Effect of Postop Steroids on Cardiovascular/Respiratory Function in Neonates Undergoing Cardiopulmonary Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jeffrey Alten, MD, Principal Investigator, Associate Professor of Pediatrics, Medical Director of the UAB Pediatric Cardiac Intensive Care Unit, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Postop Steroids after CPB
Record Dates: First submitted 2012-03-16; First posted 2012-05-10 (Estimated); Results first posted 2015-11-10 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-10

CONDITIONS: Heart Disease Congenital Complex
MeSH Terms: interventions — Hydrocortisone; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normal Saline (Placebo Comparator): The subjects will receive a bolus after successful completion of bypass and the post-pump adrenal corticotrophin hormone (ACTH) stim test equal to a 50mg/m2 dose of Hydrocortisone. This will be followed by a continuous infusion comparable to the rates a Hydrocortisone drip would run at. This infusion will be tapered down over the next 120 hours.
  Interventions: Drug: Normal Saline
- Hydrocortisone (Experimental): Subjects enrolled in this arm of the study will receive a 50mg/m2 bolus of Hydrocortisone after successful completion of CPB and the post-pump ACTH stim test has been performed. This will be followed by a continuous infusion of Hydrocortisone that will be tapered over the next 120 hours.
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Drug: Hydrocortisone — The drug will be bolused at 50mg/m2 followed by a continuous infusion that will start at 50mg/m2 for the first 48 hours and then be tapered as follows: 40mg/m2/day over 24 hours, 30mg/m2/day over 12 hours, 20 mg/m2/day over 12 hours, 10mg/m2/day over 24 hours, then off.
  Other Names: Solu Cortef
  Arms: Hydrocortisone
Drug: Normal Saline — This will be bolused and infused in the same manner as the hydrocortisone arm to ensure blinding of study arm.
  Other Names: 0.9% Sodium Chloride
  Arms: Normal Saline

SUMMARY:
This protocol is designed to offer insight into critical illness related corticosteroid insufficiency and steroid supplementation in neonates undergoing cardiac surgery with cardiopulmonary bypass by administering exogenous steroids in the immediate post-operative period.

DETAILED DESCRIPTION:
Open-heart surgery with cardiopulmonary bypass (CPB) induces an acute systemic inflammatory response (SIRS) via synthesis and release of inflammatory mediators. These inflammatory cascades may result in the development of capillary leak and generalized tissue edema, which are associated with multiorgan dysfunction involving the myocardium, lungs, kidneys, pancreas, and central nervous system. Neonates are especially susceptible to the injurious effects of SIRS. In attempt to blunt post-bypass SIRS, most neonatal heart programs have protocols in which patients receive preoperative and/or intraoperative steroids. Despite this widespread use, studies have not demonstrated consistent benefit in this therapy, and neonates often continue to suffer the deleterious effects of SIRS postoperatively. Only one study was designed to evaluate the impact of prophylactic postoperative steroid administration on outcomes after neonatal CPB. The early postoperative periods is a crucial time during which attenuation of CPB-induced SIRS by exogenous steroids may lead to improved clinical outcomes.

Adrenal insufficiency in neonates post-CPB may accentuate the harmful effects of SIRS by diminishing the anti-inflammatory and hemodynamic stabilization benefits of endogenous cortisol. Evidence suggests that neonates may suffer from inadequate cortisol activity relative to the severity of illness post-CPB, in part related to immaturity of their hypothalamic-pituitary-adrenal (HPA) axis. This so-called critical illness-related corticosteroids insufficiency (CIRCI) may contribute to low cardiac output syndrome (LCOS), respiratory dysfunction, and capillary leak in the postoperative period.

Much of the support for CIRCI as a contributor to LCOS after CPB originates from small clinical studies that demonstrate benefit of exogenous steroid supplementation on various short term clinical outcomes in patients with shock. Yet it is not clear if benefit from exogenous steroids suggests by dysregulation of the HPA axis or whether these are merely alternative effects of steroids. Investigators have recently begun to describe the cortisol response in neonates post-CPB, but there is no consensus regarding the incidence of clinically important adrenal insufficiency, its identification, or who should receive exogenous steroids.

ELIGIBILITY:
Inclusion Criteria:

1. Neonate (< 28 days old) undergoing correct cardiac surgery, or infants undergoing the following surgery procedures: Norwood, Arterial Switch, Total Anomalous Pulmonary Venous Return Repair, Interrupted Aortic Arch Repair, Truncus Arteriosus Repair
2. Successfully weaned off cardiopulmonary bypass after cardiac surgery

Exclusion Criteria:

1. requirement for extracorporeal membrane oxygenation (ECMO) in the operating room
2. Known immune deficiency
3. Having previously received systemic steroids (except for two routine preoperative doses)
4. A current signed Do not resuscitate (DNR) or limitation of care order
5. Current enrollment in another interventional clinical study
6. Refusal of parental consent
7. Previous diagnosis of adrenal insufficiency
8. > 28 days old at time of surgery whose repair dose not require CPB

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2012-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Alten, MD, Principal Investigator — UAB Pediatric Critical Care
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Saline: The subjects will receive a bolus after successful completion of bypass and the post-pump adrenocorticotrophic hormone (ACTH) stim test equal to a 50mg/m2 dose of Hydrocortisone. This will be followed by a continuous infusion comparable to the rates a Hydrocortisone drip would run at. This infusion will be tapered down over the next 120 hours.
  Normal Saline: This will be bolused and infused in the same manner as the hydrocortisone arm to ensure blinding of study arm.
- Hydrocortisone: Subjects enrolled in this arm of the study will receive a 50mg/m2 bolus of Hydrocortisone after successful completion of cardiopulmonary bypass (CPB) and the post-pump ACTH stim test has been performed. This will be followed by a continuous infusion of Hydrocortisone that will be tapered over the next 120 hours.
  Hydrocortisone: The drug will be bolused at 50mg/m2 followed by a continuous infusion that will start at 50mg/m2 for the first 48 hours and then be tapered as follows: 40mg/m2/day over 24 hours, 30mg/m2/day over 12 hours, 20 mg/m2/day over 12 hours, 10mg/m2/day over 24 hours, then off.
Period: Overall Study
Arm/Group | Normal Saline | Hydrocortisone
Started | 21 | 19
Completed | 21 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Normal Saline-Placebo: The subjects will receive a bolus after successful completion of bypass and the post-pump ACTH stim test equal to a 50mg/m2 dose of Hydrocortisone. This will be followed by a continuous infusion comparable to the rates a Hydrocortisone drip would run at. This infusion will be tapered down over the next 120 hours.
  Normal Saline: This will be bolused and infused in the same manner as the hydrocortisone arm to ensure blinding of study arm.
- Total: Total of all reporting groups
Arm/Group | Normal Saline-Placebo | Hydrocortisone | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Continuous [Median (Inter-Quartile Range); unit: Days] | 6 [5 to 11] | 5 [4 to 7] | 6 [5 to 8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 13 | 14 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 16 | 16 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 19 | 40
Surgical Procedure [Number; unit: number of patients]
  Norwood | 7 | 6 | 13
  Arterial switch operation | 6 | 6 | 12
  Interrupted aortic arch repair | 3 | 4 | 7
  Aortic arch augmentation | 1 | 1 | 2
  Truncus arteriosus repair | 3 | 0 | 3
  other | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Low Cardiac Output Syndrome (LCOS)
Description: Low Cardiac Output Syndrome (LCOS) within the first 48 hours after post-operative admission to the Pediatric Cardiac Intensive Care Unit was used as the primary outcome. This was defined as a double in inotropic support from post-operative admit, requiring Extracorporeal Membrane Oxygenation (ECMO) support, receiving Cardiopulmonary Resuscitation, or death.
Time Frame: first 48 hours after cardiac intensive care unit (CICU) admission post-op
Measure: Number; unit: percentage of patients
Arm/Group | Normal Saline-Placebo | Hydrocortisone
Number analyzed (Participants) | 21 | 19
percentage of patients | 57 | 26
Statistical Analysis 1: Comparison: Normal Saline-Placebo vs Hydrocortisone; Test type: Non-Inferiority or Equivalence — Study sample size was powered to detect a 60% difference in LCOS between groups at α 0.05 and β 0.70, assuming the prevalence of LCOS after neonatal bypass of 65% (based on retrospective data of patients who died, required rescue steroids, ECMO, or epinephrine > 0.1 μg/kg/min); p = 0.049, t-test, 2 sided — A p-value of <0.05 represents the threshold for statistical significance

2. Secondary Outcome: Mean Number of Days Subjects Alive and Ventilator Free
Description: Respiratory variables include such as alive, ventilator free days at 28 days post-op will be used as secondary outcome. The mean number of days subjects were live and ventilator free up to the 28 days after surgery.
Time Frame: up to 28 days post op
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Normal Saline-Placebo | Hydrocortisone
Number analyzed (Participants) | 21 | 19
days | 24 [17 to 26.5] | 25 [23 to 26]
Statistical Analysis 1: Comparison: Normal Saline-Placebo vs Hydrocortisone; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.44, Chi-squared

3. Secondary Outcome: Hospital Length of Stay
Description: The average length of hospital stay from the time the subject is admitted to the CICU post-op until they are discharged will be used as a secondary outcome.
Time Frame: Admit to CICU till hospital discharge, approximately 3 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Normal Saline-Placebo | Hydrocortisone
Number analyzed (Participants) | 21 | 19
days | 13.5 [9 to 24] | 19 [9 to 24]
Statistical Analysis 1: Comparison: Normal Saline-Placebo vs Hydrocortisone; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.62, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Changes in Baseline Inflammatory Mediators
Description: Changes in pre-op inflammatory mediators will be assessed at 0, 4, 12, 24 and 48 hours post bypass and used as a secondary outcome.
Time Frame: 0, 4,12, 24, and 48 hours post bypass
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Normal Saline-Placebo | Hydrocortisone
Number analyzed (Participants) | 21 | 19
pg/mL
  Pre-op Il-10 | 4 [2.9 to 5.4] | 4.3 [3 to 6.7]
  0 hr post bypass Il-10 | 225 [119 to 298] | 164 [105.3 to 312]
  4 hr post bypss Il-10 | 53.5 [31.4 to 84.9] | 92.2 [54.5 to 141]
  12 hr post bypass Il-10 | 17.5 [8.9 to 28] | 20.1 [17.3 to 34.8]
  24 hr post bypass Il-10 | 11.4 [7.9 to 21.7] | 10.7 [7 to 16.4]
  48 hr post bypass Il-10 | 7.9 [4.8 to 10.2] | 9.4 [7 to 15.4]
  Pre-op Il-1 beta | 0.49 [0.28 to 0.87] | 0.53 [0.29 to 0.78]
  0 hr post bypass Il-1 beta | 0.44 [0.28 to 1.15] | 0.5 [0.28 to 0.63]
  4 hr post bypass Il-1 beta | 0.83 [0.55 to 1.24] | 1.2 [0.58 to 1.57]
  12 hr post bypss Il-1 beta | 0.49 [0.37 to 1.37] | 0.33 [0.21 to 0.8]
  24 hr post bypass Il-1 beta | 1.71 [0.89 to 4.01] | 0.77 [0.38 to 1.13]
  48 hr post bypass Il-1 beta | 0.76 [0.45 to 1.08] | 0.29 [0.13 to 0.54]
  Pre-op Il-6 | 3.6 [1.2 to 18.8] | 5.8 [2.8 to 15.1]
  0 hr post bypass IL-6 | 13.6 [9.2 to 20.6] | 12.4 [9.7 to 19.8]
  4 hr post bypsas Il-6 | 58 [44.8 to 83.4] | 65.2 [40.3 to 89]
  12 hr post bypass Il-6 | 93.7 [61.5 to 164] | 50.4 [39.8 to 84.7]
  24 hr post bypass Il-6 | 110 [59.2 to 199] | 45.5 [33.4 to 91.6]
  48 hr post bypass Il-6 | 40.1 [23.2 to 78.9] | 15.3 [10.9 to 24.6]
  Pre-op Il-8 | 27.1 [21.7 to 37.7] | 23.5 [19.2 to 32.3]
  0 hr post bypass Il-8 | 118 [88.7 to 255] | 99.8 [71.4 to 188.5]
  4 hr post bypss IL-8 | 212 [160 to 456] | 261.5 [183.3 to 331.5]
  12 hr post bypass IL-8 | 153 [105 to 223] | 97 [62.9 to 139]
  24 hr post bypass Il-8 | 129 [97.8 to 277] | 103 [63.3 to 134.5]
  48 hr post bypass Il-8 | 67.3 [43.3 to 127] | 50.3 [37.4 to 59.1]
  Pre-op tumor necrosis factor (TNF)-alpha | 4.7 [3.4 to 5.4] | 4.3 [2.9 to 5]
  0 hr post bypass TNF-alpha | 3.6 [2.5 to 5.4] | 2.9 [2.2 to 4.1]
  4 hr post bypass TNF-alpha | 6.4 [4.5 to 8.7] | 5.5 [4.9 to 6.9]
  12 hr post bypss TNF-alpha | 6.6 [4.5 to 8.7] | 4.2 [3.2 to 4.8]
  24 hr post bypass TNF-alpha | 5.8 [4.5 to 8.7] | 4.1 [3.2 to 5]
  48 hr post bypass TNF-alpha | 5.1 [4.5 to 8.7] | 3 [2.3 to 4.4]
Statistical Analysis 1: Comparison: Normal Saline-Placebo vs Hydrocortisone; Test type: Non-Inferiority or Equivalence — There was not a power calculation for this statistic; p < 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Normal Saline-Placebo vs Hydrocortisone; Test type: Non-Inferiority or Equivalence — There was not a power calculation for this statistic; p < 0.01, Wilcoxon (Mann-Whitney) — interleukin-6 at 12, 24, and 48 hour. A p-value of <0.05 is the threshold for statistical significance
Statistical Analysis 3: Comparison: Normal Saline-Placebo vs Hydrocortisone; Test type: Non-Inferiority or Equivalence — There was not a power calculation for this statistic; p < 0.01, Wilcoxon (Mann-Whitney) — TNF-alpha at 12, 24, and 48 hours.A p-value of <0.05 is the threshold for statistical significance
Statistical Analysis 4: Comparison: Normal Saline-Placebo vs Hydrocortisone; Test type: Non-Inferiority or Equivalence — There was not a power calculation for this statistic; p < 0.05, Wilcoxon (Mann-Whitney) — Interleukin1-beta at 24 and 48 hours.A p-value of <0.05 is the threshold for statistical significance
Statistical Analysis 5: Comparison: Normal Saline-Placebo vs Hydrocortisone; Test type: Non-Inferiority or Equivalence — There was not a power calculation for this statistic; p < 0.05, Wilcoxon (Mann-Whitney) — Interleukin-8 at 24 and 48 hours.A p-value of <0.05 is the threshold for statistical significance
Statistical Analysis 6: Comparison: Normal Saline-Placebo vs Hydrocortisone; Test type: Non-Inferiority or Equivalence — There was not a power calculation for this statistic; p = 0.03, Wilcoxon (Mann-Whitney) — IL-10 at 4 hours.A p-value of <0.05 is the threshold for statistical significance

5. Secondary Outcome: Average Inotrope Score
Description: Average inotrope score over first 48 hours after Cardiac Intensive Care Unit admission was used as a secondary outcome. Inotrope Score is calculated based on the dose of inotropes currently infusing at a given time points. The formula for calculation is as follows: Epinephrine/Norepinephrine (mcg/kg/min) dose x100, plus Dopamine/Dobutamine (mcg/kg/min) dose x 1, plus Neosynephrine (mcg/kg/min) dose x10, plus Vasopressin (units/kg/hr) [(dose x60)/10,000] = Inotrope Score. Our institution does not include Milrinone in our inotrope score calculation because every patient receives a continuous infusion in the immediate post-operative period. The higher the inotrope score the more cardiac support the patient is requiring or the worse their cardiac function is becoming.
Time Frame: first 48 hours post-op
Measure: Median (Inter-Quartile Range); unit: Inotrope Score
Arm/Group | Normal Saline-Placebo | Hydrocortisone
Number analyzed (Participants) | 21 | 19
Inotrope Score
  Inotrope Score at 12 hours post bypass | 5.3 [1.5 to 12.7] | 4.7 [1.7 to 10.7]
  Inotrope Score 24 hours post bypass | 0 [0 to 7.7] | 4 [0 to 7.3]
  Inotrope Score 48 hours post bypass | 0 [0 to 7.1] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Normal Saline-Placebo vs Hydrocortisone; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p < 0.05, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Fluid Balance
Description: Hemodynamic variable such as total fluid balance within the first 48 hours post-op will be used as a secondary outcome. Fluid balance is a calculation of the overall fluid status for a given time period. The total input (fluid, medications, etc) that are given to a patient during a given time frame (24 hours) minus the total output (urine, stool, drainage, etc. ) that comes out of a patient during a given time frame.
Time Frame: 1st 48 hours post-op
Measure: Median (Inter-Quartile Range); unit: mL/kg
Arm/Group | Normal Saline-Placebo | Hydrocortisone
Number analyzed (Participants) | 21 | 19
mL/kg | -64 [-107 to 12] | -114 [-148 to -60]
Statistical Analysis 1: Comparison: Normal Saline-Placebo vs Hydrocortisone; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.04, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Changes in Baseline Arterial-venous Oxygen Saturation Difference
Description: Respiratory values such as changes in baseline arterial-venous oxygen saturation difference at admission to the pediatric cardiac intensive care unit will be used as a secondary outcome.
Time Frame: admit to the CICU
Measure: Median (Inter-Quartile Range); unit: percentage of arterial-venous saturation
Arm/Group | Normal Saline-Placebo | Hydrocortisone
Number analyzed (Participants) | 21 | 19
percentage of arterial-venous saturation | 14 [10 to 24.2] | 9.5 [7.7 to 13.5]
Statistical Analysis 1: Comparison: Normal Saline-Placebo vs Hydrocortisone; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.03, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Time Until First Extubation
Description: Respiratory values such as duration of intubation will be used as a secondary outcome.
Time Frame: Until discharge from hospital, approximately 2 weeks
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Normal Saline-Placebo | Hydrocortisone
Number analyzed (Participants) | 21 | 19
hours | 55 [21 to 195] | 51 [34 to 83]
Statistical Analysis 1: Comparison: Normal Saline-Placebo vs Hydrocortisone; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.7, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: CICU Length of Stay
Description: CICU length of stay will be calculated from the time the subject is admitted to the CICU post-op until they are discharged from the unit. This will be used as a secondary outcome.
Time Frame: approximately 1 week
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Normal Saline-Placebo | Hydrocortisone
Number analyzed (Participants) | 21 | 19
hours | 162 [137 to 389] | 213 [118 to 501]
Statistical Analysis 1: Comparison: Normal Saline-Placebo vs Hydrocortisone; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.76, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Mortality
Description: Subject mortality will in the CICU will be used as a secondary outcome.
Time Frame: Duration of CICU stay, approximately 1 week
Measure: Number; unit: percentage of patients
Arm/Group | Normal Saline-Placebo | Hydrocortisone
Number analyzed (Participants) | 21 | 19
percentage of patients | 14 | 0
Statistical Analysis 1: Comparison: Normal Saline-Placebo vs Hydrocortisone; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p = 0.23, Fisher Exact

11. Secondary Outcome: ACTH Stimulation Test
Description: AdrenoCorticoTropic Hormone stimulation test will be performed at least 24 hours pre-bypass and immediately after successful discontinuation of bypass and compared. These outcomes will be used as a secondary outcome.
Time Frame: 24 hours prebypass and 0 hours post-bypass
Measure: Median (Inter-Quartile Range); unit: microg/dL
Arm/Group | Normal Saline-Placebo | Hydrocortisone
Number analyzed (Participants) | 21 | 19
microg/dL
  Pre-op ACTH | 24.5 [10 to 33] | 31 [16.5 to 54]
  Pre-op Pre-stimulation cortisol | 18.2 [7.5 to 26] | 23.3 [11.4 to 30.4]
  Pre-op Post-stimulation cortisol | 43.6 [34.6 to 51] | 47.1 [35 to 53.3]
  Post-op ACTH | 10.5 [6.5 to 14] | 7.5 [6.4 to 9.6]
  Post-op Pre-Stimulation cortisol | 89.4 [40.5 to 130.8] | 87.2 [58.1 to 131]
  Post-op Post-stimulation cortisol | 112.3 [66.6 to 145.9] | 118.8 [72.9 to 143.4]
Statistical Analysis 1: Comparison: Normal Saline-Placebo vs Hydrocortisone; Test type: Non-Inferiority or Equivalence — Power calculations were not performed on this statistical calculation; p < 0.05, Fisher Exact
Statistical Analysis 2: Comparison: Normal Saline-Placebo vs Hydrocortisone; Test type: Non-Inferiority or Equivalence — There was not a power calculation for this statistic; p < 0.001, Fisher Exact — post-operative cortisol.A p-value of <0.05 is the threshold for statistical significance
Statistical Analysis 3: Comparison: Normal Saline-Placebo vs Hydrocortisone; Test type: Non-Inferiority or Equivalence — There was not a power calculation for this statistic; p = 0.004, Fisher Exact — Adrenal Insufficiency after bypass.A p-value of <0.05 is the threshold for statistical significance
Statistical Analysis 4: Comparison: Normal Saline-Placebo vs Hydrocortisone; Test type: Non-Inferiority or Equivalence — There was not a power calculation for this statistic; p = 0.02, Fisher Exact — Development of Low cardiac output syndrome in subjects with Adrenal Insufficiency.A p-value of <0.05 is the threshold for statistical significance

ADVERSE EVENTS:
Time Frame: Adverse events were collected from admit to the cardiac intensive care unit post-op until discharge from the cardiac intensive care unit.
Arm/Group | Normal Saline-Placebo | Hydrocortisone
Serious Adverse Events (participants affected / at risk) | 3/21 | 1/19
Other Adverse Events (participants affected / at risk) | 19/21 | 17/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Saline-Placebo (N=21) | Hydrocortisone (N=19)
Extracorporeal Membrane Oxygenation (Cardiac disorders) | 2 | 1 — Subject's requiring extracorporeal membrane oxygenation support post-cardiopulmonary bypass
Death (Surgical and medical procedures) | 3 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Saline-Placebo (N=21) | Hydrocortisone (N=19)
Acute Kidney injury (Renal and urinary disorders) | 7 | 7
Hyperglycemia (Endocrine disorders) | 15 | 10 — Subjects whose blood glucose level was >180 mg/dL
Antibiotics for suspected infection (Infections and infestations) | 8 | 7

LIMITATIONS AND CAVEATS:
small, single-center trial; included subjects from more than one surgeon; all patients received preoperative and rescue steroids; definition of low cardiac output syndrome although appropriate must ultimately be arbitrary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes